CLINICAL TRIAL: NCT06762834
Title: Investigating the Role of Ginger Tea ORAC Value in Hypertension Management
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSAHS/Batch-Spring23/023
Record Dates: First submitted 2024-12-17; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ginger Tea (Experimental)
  Interventions: Combination Product: Ginger tea
- Self Administered Tea (Active Comparator)
  Interventions: Combination Product: self administred Ginger tea

INTERVENTIONS:
Combination Product: Ginger tea — determine the optimal dosage of ginger tea that produces significant blood pressure reduction without adverse effects.
  Arms: Ginger Tea
Combination Product: self administred Ginger tea — To identify consumption and its correlation with blood pressure outcomes using a self- reported diary and periodic clinical assessments.
  Arms: Self Administered Tea

SUMMARY:
The purpose of this study is to evaluate the antihypertensive effects of ginger tea. By examining its impact on blood pressure levels, this research aims to determine whether ginger tea can be an effective, natural adjunct to conventional hypertension treatments.

DETAILED DESCRIPTION:
This investigation will provide insights into its potential role in reducing the burden of hypertension and improving cardiovascular health

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 30-65 years
* Diagnosed with stage 1 or stage 2 hypertension
* Not currently taking antihypertensive medication
* Willing to provide informed consent and adhere to study protocols.

Exclusion Criteria:

* Pregnant or breastfeeding women
* Participants on antioxidant supplements or other herbal teas.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure (SBP) | 12 Months
  Measure changes in SBP before and after the intervention with ginger tea over a defined period.
Total ORAC Value | 12 Months
  Measure the total Oxygen Radical Absorbance Capacity (ORAC) value of ginger tea consumed by participants to evaluate its antioxidant capacity and potential correlation with blood pressure changes.
Diastolic Blood Pressure (DBP) | 12 months
  Measure changes in DBP before and after the intervention with ginger tea over a defined period.

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Azra Naheed Medical College, Superior University, Lahore, Punjab Province
  - Chaudary Muhammad Akram Teaching Hospital, Azra Naheed Medical College, Superior University, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No